CLINICAL TRIAL: NCT02421484
Title: Cellular Immunotherapy for Septic Shock: A Phase I Trial
Acronym: CISS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014809
Record Dates: First submitted 2015-02-08; First posted 2015-04-20 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Septic Shock
Keywords: Phase I clinical trial; stem cell; mesenchymal stromal cell; mesenchymal stem cell
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- allogeneic mesenchymal stromal cells (Experimental): This is a Phase 1 dose escalation clinical trial that constitutes 3 dose cohorts with 3 participants per cohort who will receive intravenous doses of allogeneic bone marrow derived allogeneic mesenchymal stromal cells--0.3 million cells/kg, 1.0 million cells/kg, and 3.0 million cells/kg. We will proceed from the lower dose to the next higher dose if there are no safety concerns for each cohort.
  Interventions: Biological: Allogeneic mesenchymal stromal cells

INTERVENTIONS:
Biological: Allogeneic mesenchymal stromal cells — The allogeneic mesenchymal stromal cells will be administered intravenously.

SUMMARY:
This is a Phase I open label dose escalation trial of human allogeneic bone marrow derived mesenchymal stromal cells (MSCs) for the treatment of septic shock. The main purpose of the study is to assess the safety of MSCs in patients with septic shock.

DETAILED DESCRIPTION:
Septic shock is one of the most common and devastating health problems in the intensive care unit, with a mortality rate of approximately 40% and a staggering economic burden of approximately 4 billion dollars annually in Canada. Mesenchymal stromal cells (MSCs) may provide a promising new treatment avenue, as pre-clinical research has shown that these cells can modify a number of pathophysiological processes that are central to sepsis and greatly reduce rates of organ failure and death. This dramatic effect appears to be due to the ability of MSCs to modify the inflammatory cascade, augment tissue repair and enhance pathogen clearance. MSCs have been evaluated in randomized clinical trials including those with myocardial infarction, heart failure, neurological and metabolic disorders, hematological malignancies, and chronic obstructive pulmonary disease with no serious safety concerns. However, MSC therapy has not yet been evaluated in humans with septic shock. Prior to a randomized controlled trial to examine the efficacy of MSCs in septic shock, an evaluation of safety is necessary. The Cellular Immunotherapy for Septic Shock (CISS) trial is an open label Phase I dose escalation trial that will evaluate the safety of MSC therapy in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all 5 inclusion criteria to be eligible:

1. Admission to the Ottawa Hospital Intensive Care Unit
2. Receipt of appropriate broad spectrum antibiotics for the suspected/confirmed infectious source and adequate source control according to the opinion of the treating critical care physician
3. Within 24 hours of admission to the ICU, receipt of reasonable levels of fluid administration and resuscitation as indicated by:

   * a central venous pressure of at least 8 mm Hg AND
   * a central venous oxygen saturation of at least 70%.
4. Cardiovascular failure that is present within the first 24 hours of admission to the ICU and that is present for at least 4 consecutive hours AND
5. Deterioration or lack of improvement in at least 1 additional organ function, or organ hypoperfusion, as defined by the modified Multiple Organ Dysfunction Score (MODS). Criteria for organ dysfunction or organ hypoperfusion must be met within the first 24 hours of ICU admission

Exclusion Criteria:

1. Another form of shock (cardiogenic, hypovolemic, obstructive) that is considered by the treating critical care physician as the dominant cause of shock
2. History of known pulmonary hypertension with a WHO functional class of III or IV
3. History of severe pulmonary disease requiring home oxygen
4. History of severe cardiac disease with a New York Heart Association Functional Class of III or IV, or severe ischemic heart disease with a Canadian Cardiovascular Society angina class score of III or IV
5. History of severe liver disease (Child class C)
6. Malignancy in the previous 2 years (excluding resolved non-melanoma skin cancer).
7. Chronic immune suppression
8. History of anaphylaxis
9. Pregnant or lactating
10. Enrolment in another interventional study
11. Family, participant, or physician not committed to aggressive care
12. Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | 12 months
  A historical cohort that met CISS eligibility criteria were previously enrolled to compare the incidence of adverse events with the CISS interventional arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lauralyn McIntyre, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The sample size of the interventional arm is very small and the sharing of individual data has privacy and confidentiality implications.

REFERENCES:
- [Derived] McIntyre LA, Stewart DJ, Mei SHJ, Courtman D, Watpool I, Granton J, Marshall J, Dos Santos C, Walley KR, Winston BW, Schlosser K, Fergusson DA; Canadian Critical Care Trials Group; Canadian Critical Care Translational Biology Group. Cellular Immunotherapy for Septic Shock. A Phase I Clinical Trial. Am J Respir Crit Care Med. 2018 Feb 1;197(3):337-347. doi: 10.1164/rccm.201705-1006OC. PMID 28960096